CLINICAL TRIAL: NCT06356818
Title: Comparison of Virtual Reality and Motor Imagery Applications in Patients With Ankle Instability
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Doaa Tarek Fathy Elsayed HAKAM, Physiotherapist, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-74555795-050.04-941155
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Ankle Sprains
Keywords: Ankle instability; Virtual reality (VR); Motor imagery (MI); Rehabilitation technology
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Intervention Model Description: three groups with a conventional therapy control group.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional physiotherapy program group (Active Comparator): Physiotherapy and rehabilitation treatment program will be applied to the patients. In this program, a 30-40-minute exercise protocol including proprioceptive, balance and strengthening exercises will be applied.
  Interventions: Other: Conventional physiotherapy program
- Virtual reality (VR) program group (Active Comparator): Virtual reality (VR) program will be applied in addition to the conventional physiotherapy program. In VR; the subjects will be asked to stand on the Wii fit balance board and will be able to physically and visually see and participate in the game. Nintendo Wii Fit Plus will last 30 minutes in total as warm-up exercise (5 minutes), workout (20 minutes) and cool-down exercise (5 minutes). Interactive video games will be used, including both strength and balance exercises. The exercises in the study include 5 muscle strengthening (e.g. forward lunge/ lunge, single leg extension, side leg raise, single leg bend, rowing) and 5 balance exercises (e.g. playing soccer, ski slalom, tightrope walk, snowboard slalom) among the programs built into the Nintendo Wii Fit Plus.
  Interventions: Other: Conventional physiotherapy program; Other: Virtual reality (VR)
- Motor imagery (MI) program group (Active Comparator): In addition to VR and conventional physiotherapy programs motor imagery program will be given to the patients in this group. Using the explicit MI method, individuals will be explicitly instructed to perform imagery (2). The physiotherapist will ask the patient to imagine a real or fantasy place that is peaceful, happy and relaxing. Then, they will be asked to imagine that they are in this picture. Patients will be asked to imagine themselves doing physiotherapy exercises and feel the movements as vividly as possible. The content of the imagery program will last 20 minutes in total, with 5 minutes of relaxation and 15 minutes of imagery training.
  Interventions: Other: Conventional physiotherapy program; Other: Virtual reality (VR); Other: Motor imagery (MI)

INTERVENTIONS:
Other: Conventional physiotherapy program — Physiotherapy and rehabilitation treatment program will be applied to the patients. In this program, a 30-40-minute exercise protocol covering proprioceptive, balance and strengthening exercises will be implemented. For a total of 12 sessions, 3 days a week, over a 4-week period
Other: Virtual reality (VR) — virtual reality (VR) program will be applied using balance and strengthening games by Nintendo Wii Fit Plus; warm-up exercise (5 minutes), workout (20 minutes) and cool-down exercise (5 minutes) for a total of 30 minutes. For a total of 12 sessions, 3 days a week, over a 4-week period
  Arms: Motor imagery (MI) program group; Virtual reality (VR) program group
Other: Motor imagery (MI) — Patients will be introduced to explicit Motor imagery program which the content of the imagery program will last 20 minutes in total, with 5 minutes of relaxation and 15 minutes of imagery training. For a total of 12 sessions, 3 days a week, over a 4-week period.
  Arms: Motor imagery (MI) program group

SUMMARY:
In this study, the effects of different treatment methods for ankle instability patients are being compared aiming to find the optimal treatment. Via comparing virtual reality, motor imagery, and classic rehabilitation programs to clarify their effects on ankle static and dynamic balance, proprioception, range of motion, muscle strength, pain, function and patient satisfaction.

DETAILED DESCRIPTION:
This study will be carried out at Istanbul University-Cerrahpaşa Department of Physiotherapy and Rehabilitation with 30 participants. Subjects who meet the inclusion criteria and who voluntarily agree to participate in this study will be randomly divided into 3 study groups as conventional physiotherapy rehabilitation treatment program, Conventional + virtual reality (VR) group and Conventional + VR+ motor imagery (MI) group. Group 1 (Conventional physiotherapy program): Physiotherapy and rehabilitation treatment program will be applied to the patients. In this program, a 30-40-minute exercise protocol covering proprioceptive, balance and strengthening exercises will be implemented. Group 2; VR group: in addition to the conventional physiotherapy program virtual reality (VR) program will be applied to this group using balance and strengthening games by Nintendo Wii Fit Plus; warm-up exercise (5 minutes), workout (20 minutes) and cool-down exercise (5 minutes) for a total of 30 minutes. Group 3; Motor imagery (MI): this group will be introduced to explicit Motor imagery program adding to Conventional physiotherapy and VR programs. The content of the imagery program will last 20 minutes in total, with 5 minutes of relaxation and 15 minutes of imagery training.

All patients in the groups will be treated for a total of 12 sessions, 3 days a week, over a 4-week period. Session duration will vary according to the groups. Interventions will last approximately 40-80 minutes.

Ankle mobility and instability will be assessed through different tests. Balance parameters will be measured with the Star Balance Test for dynamic balance and the Single Leg Stance Test for static balance. The pain intensity will be measured with the Pressure Pain Threshold device also with Visual Analog Scale. Muscle strength will be assessed with a manual muscle test. Ankle range of motion and joint position feeling will be measured with a mobile application such as an inclinometer. Finally, 2 questionnaires will be used to assess functional ability and patient satisfaction. These are; Cumberland ankle instability tool and Global Assessment Scale questionnaire respectively. All of the assessment parameters (outcomes measurement) will be evaluated twice, pre-treatment and post-treatment (after 4 weeks).Which approximately will take from 30 to 45 minutes.

G*Power analysis program was used to calculate the sample size of the study. While the Cumberland ankle instability tool (CAIT) change results were taken as reference, the effect size was calculated as 1.35, and the number of subjects to be included in the study was reported as a total of 15 patients (Group 1: 5/Group 2: 5/Group 3: 5) in order to be determined as significant with 95% power and type 1 error=0.05,however, the exclusion rate was added as 25% and it has been decided to include a total of 30 patients (Group 1: 10/Group 2: 10/Group 3: 10) (1). SPSS (Statistical Package for Social Sciences) (SPSS 20.0) statistical program will be used for statistical analysis of the data obtained. In all analyzes, p<0.05 will be considered statistically significant. Before the final analysis, the data will be screened to test the normality assumption using the Shapiro-Wilk test, which reflects normal distribution (p > 0.05). Furthermore, Levene's test was used to test homogeneity of variance and no significant difference was found (p > 0.05). If the data are normally distributed, parametric analysis (e.g. t-Test, ANOVA, Paired t-Test and Linear Regression) will be used, otherwise non-parametric analysis (e.g. Mann-Whitney U Test, Wilcoxon Signed-Rank Test, Kruskal-Wallis Test and Spearman's Rank Correlation) will be used.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with ≤27 points according to the Cumberland ankle parameter (≤27 points represent unstable ankles) (12).
* Patients with both mechanical and functional instability
* Patients with instability after ankle sprain
* Patients with sub-acute (10 days after injury) and chronic ankle instability
* Diseases/patients without surgical indication
* Cases between the ages of 18-39
* Gender (Male-Female)

Exclusion Criteria:

* Patients with acute ankle instability
* Athletes with ankle instability
* Previous history of lower extremity surgery
* Those with a Cumberland Ankle Instability Instrument (CAIT) score of less than 24.
* Cannot walk without a supportive walking aid.
* Participants in another exercise program that may affect their feet.
* Subjects who have been involved in different treatments for instability in the last 3 months
* Patients with neurologic, rheumatologic or vestibular problems will be excluded (14).

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | two weeks
  Visual Analog Scale (VAS) will be used for pain assessment. This test is a subjective, valid, and reliable test also it is time-saving and easy to apply and understand by the patient as the patient will be asked to scale their pain from 0 to 10 as 0 referring to: no pain and 10 referring to : maximum severe pain.
Pressure Pain Threshold (PPT) | two weeks
  The Pressure Pain Threshold (PPT) is used to measure pain. This test is an objective valid, and reliable test which will provide us with more accurate results according to the sensation of pain. It is also time-saving and easy to apply. The PPT test will be applied to the most painful area on the ankle joint and the result will be compared with the other extremity, as well as with a healthy area close to an area such as the tibialis anterior. The calculation will be done with kilograms.
Star Excursion Balance Test (SEBT) | two weeks
  Dynamic balance and instability will be evaluated using the Star Excursion Balance Test (SEBT) for dynamic balance assessment. This test is time-efficient and does not require the use of special equipment. It could be proceeded easily with a simple setup four strips of tape will need to be cut to a length of 183 to 244 cm each. Two pieces will be used to form a '+', with the other two being placed over top to form an 'x' so that a star shape is formed. It is important that all lines are separated from each other by a 45° angle. The goal of the SEBT is to maintain a single leg stance on one leg while reaching as far as possible with the contralateral leg. The results will be obtained in centimeters.
Single Leg Balance Test (SLBT) | two weeks
  The Single Leg Balance Test (SLBT) will be used to assist static balance. This test is applicable easy test without any need for special devices or setup. Simply we will ask the participant to stand on one leg and we will calculate the average of three trials in each limb, the patient will be administered for 3 minutes with eyes open and another 3 minutes with eyes closed with a maximum time of one minute for each trial. The duration starts when the patient lifts his foot off the ground and ends when his foot touches the ground. The test ends when the foot moves, or the time reaches the maximum (60 seconds).
Joint position sense (JPS) | two weeks
  Proprioception, Joint position sense (JPS) will be measured using mobile applications such as Tiltmeter for iPhone and Handy Level (inclinometer) for Android (8). Nowadays using mobile applications for assessment is becoming a widely accepted, valid and reliable method which is affordable and applicable. In order to accurately calculate JPS the active ankle repositioning technique will be used. Individuals will be asked to relocate their feet in dorsiflexion and plantarflexion directions to two targets (10° and 15°). During the JPS measurements, all patients will be blindfolded to eliminate the contribution of vision.
Range of Motion (ROM) | two weeks
  Range of Motion (ROM), will be calculated with inclinometer mobile application. Using mobile application will make it easier to obtain ankle ROM (dorsiflexion, planterflexion, inversion and eversion). In this test ROM will be calculated to clarify the baseline (normal range of motion) of the ankle and find out the changes before and after the intervention. Also to perform the proprioception test from the correct starting position.
Muscle strength | two weeks
  Lower extremity muscle strength will be assessed using manual muscle testing (MMT). MMT is a fundamental method which is not requiring any devices or setup. We will use the available literature as a reference to apply MMT in the most reliable and valid way. According to the evaluation method (0 - No contraction, 1 - Vibration or feeling of contraction, 2 - Active movement with removal of gravity, 3 - Active movement against gravity, 4 - Active movement against gravity and resistance, 5 - Normal strength) (10). Plantarflexors, dorsiflexors muscle groups, tibialis anterior muscle and hip abductor muscle group will be evaluated.

SECONDARY OUTCOMES:
Cumberland ankle instability questionnaire (CAIT) | two weeks
  Functional ability will be assessed with the Cumberland ankle instability questionnaire (CAIT). Which is a valid, reliable, time-saving and easily understood tool. The CAIT is a 9-item 30-point scale using a numeric value that measures the severity of ankle instability. The participant will be asked to answer these questions for both ankles.
Patient satisfaction | two weeks
  By using the Global Rating Scale patient satisfaction will be measured by asking the patient directly how satisfied they are with the treatment provided. This tool is an easy direct one ,which is a 5-point Likert scale. Patient Satisfaction (after treatment) is scored as: much worse, worse, same, better and much better.

CONTACTS AND LOCATIONS:
Overall Officials: YILDIZ AKBABA, Assoc. Prof., Principal Investigator — Istanbul University - Cerrahpasa; Doaa HAKAM, PT, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa (IUC), Istanbul, Turkey (Türkiye)